CLINICAL TRIAL: NCT02958514
Title: Efficacy Comparison of Two Kinds of Treatment in Treating Dry Eye Caused by Meibomian Gland Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Hong Qi, MD.PHD., Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016154
Record Dates: First submitted 2016-10-03; First posted 2016-11-08 (Estimated); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Dry Eye Syndrome
Keywords: IPL; MGD
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Intense Pulsed Light Therapy; Tobramycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- traditional treatment group (Other): Subjects in this group are treated by tobramycin and dexamethasone ophthalmic ointment qn and artificial tears qid.
  Interventions: Drug: Tobramycin and Dexamethasone Ophthalmic Ointment
- IPL treatment group (Experimental): Subjects in this group are treated with 3 cycles of intense pulsed light of 4 weeks interval and artificial tears qid.
  Interventions: Device: intense pulsed light

INTERVENTIONS:
Device: intense pulsed light — Intense pulse light (IPL) has been used in dermatology practices for several years as a treatment for rosacea and acne.IPL uses Xenon flashlamp to emit wavelengths of light from 400 to 1200nm. When placed on the light, a filter restricts the wavelength to the visible light range of *500nm.In 2007-2008, an IPL treatment technology-the Diamond Q4 by DermaMed Solutions-was specifically configured to our specifications with the goal of stimulating secretion of normal meibum via skin treatment effects on the meibomian glands. It was discovered that dry eye patients are better positioned for gland expression, as IPL seems to liquefy the abnormal viscous meibum and dilate the glands.
  Arms: IPL treatment group
Drug: Tobramycin and Dexamethasone Ophthalmic Ointment
  Arms: traditional treatment group

SUMMARY:
This study aims to evaluate the efficacy of intense pulsed light in treating dry eye caused by meibomian gland dysfunction and make a comparison between the traditional treatment.

ELIGIBILITY:
Inclusion Criteria:

* patients with dry eye syndrome and diagnosed as MGD

Exclusion Criteria:

* an infection or inflammatory disease;
* ocular surgical history with in the last 3 months
* SGOGREN SYNDROME

Ages: 26 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Ocular Surface Disease Index (OSDI) | through study completion,an average of 6 months
  normal value：<13 abnormal value：≥ 13

SECONDARY OUTCOMES:
The concentrations of inflammatory cytokines such as IL-1、IL-6 and IL-8 | through study completion,an average of 6 months
breakup time of tear film （BUT） | through study completion,an average of 6 months
  normal value：>10s abnormal value：≤ 10s
Corneal Fluorescein Stain(CFS) | through study completion,an average of 6 months
Eyelid ester discharge ability score | through study completion,an average of 6 months
Eyelid ester trait ratings | through study completion,an average of 6 months

IPD SHARING:
Plan to Share IPD: Yes